CLINICAL TRIAL: NCT03354273
Title: A Phase 3, Open-Label, Multicentre Study of Flurpiridaz (18F) Injection for Positron Emission Tomography (PET) Imaging for Assessment of Myocardial Perfusion in Patients Referred for Invasive Coronary Angiography Because of Suspected Coronary Artery Disease
Brief Title: An International Study to Evaluate Diagnostic Efficacy of Flurpiridaz (18F) Injection PET MPI in the Detection of Coronary Artery Disease (CAD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: Pharmaceutical Product Development, (PPD) LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-265-303; 2017-005011-14 (EudraCT Number)
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Results first posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-06

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: Positron emission tomography myocardial perfusion imaging (PET MPI); Single photon emission computed tomography myocardial perfusion imaging (SPECT MPI); Invasive coronary angiography (ICA); Coronary artery disease (CAD)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Flurpiridaz PET MPI (following off-study SPECT MPI)
  Interventions: Drug: PET MPI; Drug: SPECT MPI; Drug: Pharmacological stress agents

INTERVENTIONS:
Drug: PET MPI — Flurpiridaz (18F) Injection. All participants received 2 IV boluses of Flurpiridaz (18F) Injection in a large peripheral vein: 1 at rest and 1 during stress. The dosages of Flurpiridaz (18F) Injection administered at rest and during stress conditions did not exceed a total of 14 mCi (520 MBq) for an individual participant.
Drug: SPECT MPI — SPECT imaging was used 99mTc-based myocardial tracers. SPECT agents utilised for the purposes of this clinical study was administered as per American Society of Nuclear Cardiology or European Association of Cardiovascular Imaging standards, where applicable. All participants undergone SPECT MPI.
Drug: Pharmacological stress agents — Pharmacologic stress agents were restricted to the following 3 agents, as permitted by local marketing authorisations and availability: adenosine, dipyridamole, and regadenoson. Administration was through an IV line.

SUMMARY:
This is a Phase 3, prospective, open-label, international, multicentre study of Flurpiridaz (18F) Injection for PET MPI in patients referred for ICA because of suspected CAD.

ELIGIBILITY:
Inclusion Criteria:

* The participant was a man or woman ≥18 years of age.
* The participant had read, signed, and dated an informed consent form (ICF) prior to any study procedures being performed.
* At the time of enrolment, the participant had been scheduled via written documentation to undergo an ICA for the assessment of CAD.
* The participant had undergone a clinically indicated SPECT OR the participant was willing to undergo SPECT MPI for the purposes of the clinical study.
* The participant was male or was a nonpregnant, nonlactating female who was either surgically sterile or was post-menopausal.
* The participant was able and willing to comply with all study procedures as described in the protocol.

Exclusion Criteria:

* Participants who were pregnant, may possibly be pregnant, or wish (including their partners) to became pregnant during the study period, or were lactating.
* Participants who were unable to undergo all of the imaging procedures.
* Participants who had an established diagnosis of CAD as confirmed by any of the following:

  1. Previous myocardial infarction (MI);
  2. Previous cardiac catheter angiography showing ≥50% stenosis;
  3. Previous coronary revascularisation, such as percutaneous coronary intervention (PCI), thrombolysis or coronary artery bypass graft (CABG) placement.
* Participants incapable of undergoing either exercise or pharmacological cardiac stress testing.
* Participants who had a current illness or pathology that, in the opinion of the investigator, would pose a significant safety risk for the participant during cardiac stress testing.
* Documented history of heart failure and/or cardiomyopathy and/or prior LV ejection fraction (LVEF) <50%).
* Participants scheduled for or planning to undergo any cardiac interventional procedures between enrolment and ICA.
* Participants undergoing evaluation for heart transplantation or with history of heart transplantation.
* Participants enrolled in another clinical study within the 30 days prior to being enrolled in this study or scheduled to participate in another clinical study during the 7-day follow-up period of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francois Tranquart, M.D., Ph.D., Study Director — General Electric Healthcare Life Sciences
Locations (53):
- United States (37):
  - Vascular Biology and Hypertension Program, University of Alabama at Birmingham, Birmingham, Alabama
  - University of California- Los Angeles, Los Angeles, California
  - Keck Hospital of USC, Los Angeles, California
  - VA Greater Los Angeles Health Care System, Los Angeles, California
  - VA San Diego Health System, San Diego, California
  - UCSF, San Francisco, California
  - Tower Saint John's Imaging, Santa Monica, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Cardiology Physicians PA/Red Clay Research LLC, Newark, Delaware
  - University of Florida, Gainesville, Florida
  - Indago Research and Health Center, Hialeah, Florida
  - Optimus U Corp, Miami, Florida
  - Infinite Clinical Research, Miami, Florida
  - Allied Biomedical Research Institute, Miami, Florida
  - Comprehensive Vascular Care PA, Miami, Florida
  - Amavita Clinical Research, LLC, North Miami Beach, Florida
  - Emory University, Atlanta, Georgia
  - University Of Iowa Hospitals And Clinics, Iowa City, Iowa
  - Midwest Heart and Vascular Specialists, Overland Park, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - VA St. Louis Health Care System, St Louis, Missouri
  - St Louis University, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center/New York Presbyterian Hospital - Milstein Hospital Building, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Berks Cardiologists, LTD, Wyomissing, Pennsylvania
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - VA North Texas Health Care System - NAVREF - PPDS, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - Vital Heart & Vein, Humble, Texas
  - Memorial City and Katy Cardiology Associates, Katy, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Roanoke Heart Institute, Roanoke, Virginia
- Canada (3):
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Center Hospitalier Universitaire de Sherbrooke CHUS, Montreal, Quebec
- Turku University Hospital, Turku, Finland
- France (3):
  - Hopital Cote de Nacre, Caen
  - Groupe Hospitalier Bichat Claude Bernard, Paris
  - Centre Cardiologique Du Nord, Saint-Denis
- Germany (2):
  - Universitätsklinikum der RWTH Aachen, Aachen
  - Universitätsklinikum Essen, Essen
- Netherlands (5):
  - VU Medisch Centrum, Amsterdam
  - Amphia Ziekenhuis - WCN - PPDS, Breda
  - Catharina Hospital, Eindhoven
  - Zuyderland Medisch Centrum-WCN-PPDS, Heerlen
  - Leids Universitair Medisch Centrum, Leiden
- Switzerland (2):
  - Hopitaux Universitaires de Geneve, Geneva
  - Universitatsspital Zurich, Zurich

REFERENCES:
- [Derived] Maddahi J, Agostini D, Bateman TM, Bax JJ, Beanlands RSB, Berman DS, Dorbala S, Garcia EV, Feldman J, Heller GV, Knuuti JM, Martinez-Clark P, Pelletier-Galarneau M, Shepple B, Tamaki N, Tranquart F, Udelson JE. Flurpiridaz F-18 PET Myocardial Perfusion Imaging in Patients With Suspected Coronary Artery Disease. J Am Coll Cardiol. 2023 Oct 17;82(16):1598-1610. doi: 10.1016/j.jacc.2023.08.016. PMID 37821170
- [Derived] Bourque JM, Hanson CA, Agostini D, Bateman TM, Bax JJ, Beanlands RSB, Berman DS, Garcia EV, Heller GV, Knuuti J, Tamaki N, Udelson JE, Maddahi J. Assessing myocardial perfusion in suspected coronary artery disease: rationale and design of the second phase 3, open-label multi-center study of flurpiridaz (F-18) injection for positron emission tomography (PET) imaging. J Nucl Cardiol. 2021 Jun;28(3):1105-1116. doi: 10.1007/s12350-021-02527-8. Epub 2021 Jan 31. PMID 33521873

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 48 centers in Finland, France, Germany, Netherlands, United States and Canada from 05 June 2018 to 05 May 2022.
Pre-assignment Details: A total 730 participants signed informed consent and were enrolled, of these, 604 participants received greater than or equal to (>=) 1 dose of Flurpiridaz (18F) Injection in this study.
Groups:
- Flurpiridaz (18F): All Participants: Participants received 2 intravenous (IV) boluses of Flurpiridaz (18F) Injection in a large peripheral vein: 1 at rest then 1 during stress on the same day within 60 days prior to the invasive coronary angiography (ICA). Flurpiridaz (18F) Injection administered at rest and during stress conditions were not to exceed a total of 14 millicurie (mCi) (520 megabecquerel [MBq]) for an individual participant. Flurpiridaz was administered on Study Day 1.
  Single photon emission computed tomography (SPECT) agents 99mTc-based myocardial tracers, example [99mTc]tetrofosmin or [99mTc]sestamibi were administered as per American Society of Nuclear Cardiology or European Association of Cardiovascular Imaging standards corresponding to study site location. For each participant, the same stress type (pharmacologic or exercise) was used for the SPECT and Flurpiridaz (18F) Injection positron emission tomography (PET) myocardial perfusion imaging (MPI). Also, if pharmacological stress was used, the same agent and the same dose of pharmacological stress agent was used for both types of imaging for the same participant.
  Pharmacological stress agents were administered according to the respective Package Insert (as applicable) or American Society of Nuclear Cardiology or European Association of Cardiovascular Imaging standards corresponding to study site location.
Period: Overall Study
Arm/Group | Flurpiridaz (18F): All Participants
Started | 730 (Participants who signed informed consent form and were enrolled in the study.)
Safety Population (Treated) | 604
Modified Intent-to-Treat (MITT) Population | 578
Secondary Modified Intent-to-Treat (SMITT) Population | 578
Completed | 578
Not Completed | 152
Not completed — Adverse Event | 5
Not completed — Screen Failure | 21
Not completed — Withdrawal by Subject | 34
Not completed — Technical Problems | 30
Not completed — Lost to Follow-up | 4
Not completed — Investigator Decision | 3
Not completed — Investigational Medicinal Product (IMP) Supply Issues | 21
Not completed — Issues With Performing Invasive Coronary Angiography (ICA) | 20
Not completed — COVID-19 Restrictions | 9
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Population: The enrolled population consisted of all participants who signed informed consent.
Groups:
- Flurpiridaz (18F): All Participants: Participants received 2 IV boluses of Flurpiridaz (18F) Injection in a large peripheral vein: 1 at rest then 1 during stress on the same day within 60 days prior to the ICA. Flurpiridaz (18F) Injection administered at rest and during stress conditions were not to exceed a total of 14 mCi (520 MBq) for an individual participant. Flurpiridaz was administered on Study Day 1.
  SPECT agents 99mTc-based myocardial tracers, example [99mTc]tetrofosmin or [99mTc]sestamibi were administered as per American Society of Nuclear Cardiology or European Association of Cardiovascular Imaging standards corresponding to study site location. For each participant, the same stress type (pharmacologic or exercise) was used for the SPECT and Flurpiridaz (18F) Injection PET MPI. Also, if pharmacological stress was used, the same agent and the same dose of pharmacological stress agent was used for both types of imaging for the same participant.
  Pharmacological stress agents were administered according to the respective Package Insert (as applicable) or American Society of Nuclear Cardiology or European Association of Cardiovascular Imaging standards corresponding to study site location.
Arm/Group | Flurpiridaz (18F): All Participants
Number analyzed (Participants) | 730
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (9.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 235
  Male | 495
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 98
  Not Hispanic or Latino | 512
  Unknown or Not Reported | 120
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 55
  White | 579
  More than one race | 0
  Unknown or Not Reported | 82
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 129
  United States | 412
  Finland | 36
  France | 71
  Germany | 3
  Netherlands | 79

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of Flurpiridaz (18F) Injection Positron Emission Tomography (PET) Myocardial Perfusion Imaging (MPI) in the Detection of Significant Coronary Artery Disease (CAD) as Defined by Cardiac Catheterization
Description: Sensitivity was defined as true positives (TP)/(TP+false negatives [FN]). TP was participants with abnormal PET MPI and disease positive by truth standard and FN was participants with normal PET MPI and disease positive by truth standard. Specificity defined as true negatives (TN)/(TN+ false positives [FP]). TN was participants with normal PET MPI and disease negative by truth standard and FP was participants with abnormal PET MPI and disease negative by truth standard. Truth standard was presence of CAD as evidenced by presence of stenosis of >=50 percent (%) in >=1 coronary artery or major branch of a coronary artery as determined by quantitative coronary angiography (QCA) analysis. Participants were considered to have CAD if QCA revealed >=50% stenosis of >=1 major coronary artery or major branch. Sensitivity and specificity were calculated for 3 readers and majority rule using each participant judgement (positive or negative) by at least 2 of 3 readers.
Time Frame: Up to 60 days
Population: The MITT population included all participants who completed the rest and stress Flurpiridaz (18F) Injection PET MPI procedures and who had evaluable truth standard data. Here, "overall number of participants analyzed" signifies participants who were analyzed for a specific reader (combined sensitivity or specificity) and "number analyzed" signifies participants who were evaluable for specified categories.
Measure: Number (95% Confidence Interval); unit: percent
Groups:
- Flurpiridaz (18F): Participants received 2 IV boluses of Flurpiridaz (18F) Injection in a large peripheral vein: 1 at rest then 1 during stress on the same day within 60 days prior to the ICA. Flurpiridaz (18F) Injection administered at rest and during stress conditions were not to exceed a total of 14 mCi (520 MBq) for an individual participant. Flurpiridaz was administered on Study Day 1.
  SPECT agents 99mTc-based myocardial tracers, example [99mTc]tetrofosmin or [99mTc]sestamibi were administered as per American Society of Nuclear Cardiology or European Association of Cardiovascular Imaging standards corresponding to study site location. For each participant, the same stress type (pharmacologic or exercise) was used for the SPECT and Flurpiridaz (18F) Injection PET MPI. Also, if pharmacological stress was used, the same agent and the same dose of pharmacological stress agent was used for both types of imaging for the same participant.
  Pharmacological stress agents were administered according to the respective Package Insert (as applicable) or American Society of Nuclear Cardiology or European Association of Cardiovascular Imaging standards corresponding to study site location.
Arm/Group | Flurpiridaz (18F)
Number analyzed (Participants) | 578
percent
  Reader 1: Sensitivity: number analyzed (Participants) | 249
  Reader 1: Sensitivity | 77.1 [71.9 to 82.3]
  Reader 1: Specificity: number analyzed (Participants) | 329
  Reader 1: Specificity | 65.7 [60.5 to 70.8]
  Reader 2: Sensitivity: number analyzed (Participants) | 249
  Reader 2: Sensitivity | 73.5 [68.0 to 79.0]
  Reader 2: Specificity: number analyzed (Participants) | 329
  Reader 2: Specificity | 69.6 [64.6 to 74.6]
  Reader 3: Sensitivity: number analyzed (Participants) | 249
  Reader 3: Sensitivity | 88.8 [84.8 to 92.7]
  Reader 3: Specificity: number analyzed (Participants) | 329
  Reader 3: Specificity | 52.6 [47.2 to 58.0]
  Majority Rule: Sensitivity: number analyzed (Participants) | 249
  Majority Rule: Sensitivity | 80.3 [75.4 to 85.3]
  Majority Rule: Specificity: number analyzed (Participants) | 329
  Majority Rule: Specificity | 63.8 [58.6 to 69.0]
Statistical Analysis 1: Comparison: Flurpiridaz (18F); Reader 1: Sensitivity; Test type: Other — Sensitivity was compared to a pre-specified threshold of 60%; p < 0.0001, One-sided z-tests; The hypothesis tests were one-sided z-tests with a significance level of 0.025
Statistical Analysis 2: Comparison: Flurpiridaz (18F); Reader 1: Specificity; Test type: Other — Specificity was compared to a pre-specified threshold of 60%; p = 0.0182, One-sided z-tests; The hypothesis tests were one-sided z-tests with a significance level of 0.025
Statistical Analysis 3: Comparison: Flurpiridaz (18F); Reader 2: Sensitivity; Test type: Other — Sensitivity was compared to a pre-specified threshold of 60%; p < 0.0001, One-sided z-tests; The hypothesis tests were one-sided z-tests with a significance level of 0.025
Statistical Analysis 4: Comparison: Flurpiridaz (18F); Reader 2: Specificity; Test type: Other — Specificity was compared to a pre-specified threshold of 60%; p = 0.0002, One-sided z-tests; The hypothesis tests were one-sided z-tests with a significance level of 0.025
Statistical Analysis 5: Comparison: Flurpiridaz (18F); Reader 3: Sensitivity; Test type: Other — Sensitivity was compared to a pre-specified threshold of 60%; p < 0.0001, One-sided z-tests; The hypothesis tests were one-sided z-tests with a significance level of 0.025
Statistical Analysis 6: Comparison: Flurpiridaz (18F); Reader 3: Specificity; Test type: Other — Specificity was compared to a pre-specified threshold of 60%; p = 0.9970, One-sided z-tests; The hypothesis tests were one-sided z-tests with a significance level of 0.025
Statistical Analysis 7: Comparison: Flurpiridaz (18F); Majority Rule: Sensitivity; Test type: Other — Sensitivity was compared to a pre-specified threshold of 60%; p < 0.0001, One-sided z-tests; The hypothesis tests were one-sided z-tests with a significance level of 0.025
Statistical Analysis 8: Comparison: Flurpiridaz (18F); Majority Rule: Specificity; Test type: Other — Specificity was compared to a pre-specified threshold of 60%; p = 0.0781, One-sided z-tests; The hypothesis tests were one-sided z-tests with a significance level of 0.025

2. Secondary Outcome: Sensitivity and Specificity of Flurpiridaz (18F) Injection PET MPI Compared SPECT MPI for All Participants When the Diagnosis of CAD by ICA Was the Standard of Truth
Description: Sensitivity:TP/(TP+FN). TP:participants with abnormal PET MPI and disease positive by truth standard and FN:participants with normal PET MPI and disease positive by truth standard. Specificity:TN/(TN+ FP). TN:participants with normal PET MPI and disease negative by truth standard and FP:participants with abnormal PET MPI and disease negative by truth standard. Truth standard was presence of CAD as evidenced by presence of stenosis of >=50% in >=1 coronary artery or major branch of coronary artery as determined by QCA analysis. Participants considered to have CAD if QCA revealed >=50% stenosis of >=1 major coronary artery or major branch. Sensitivity, specificity was calculated for 3 readers and majority rule using each participant judgement (positive or negative) by at least 2 of 3 readers. Sensitivity, specificity of Flurpiridaz (18F) PET MPI compared to SPECT MPI with QCA as standard of truth at >=50% stenosis threshold for all participants was reported by reader and majority rule.
Time Frame: Up to 60 days
Population: The SMITT population included the participants who completed the rest and stress SPECT MPI (if the participant's SPECT MPI was "off-study," that SPECT MPI had to meet minimal quality standards, as specified by the imaging core lab). Here, "overall number of participants analyzed" signifies participants who were analyzed for a specific reader (combined sensitivity or specificity) and "number analyzed" signifies participants who were evaluable for specified categories.
Measure: Number (95% Confidence Interval); unit: percent
Groups:
- Flurpiridaz (18F) PET MPI: Participants received 2 IV boluses of Flurpiridaz (18F) Injection in a large peripheral vein: 1 at rest then 1 during stress on the same day within 60 days prior to the ICA. Flurpiridaz (18F) Injection administered at rest and during stress conditions were not to exceed a total of 14 mCi (520 MBq) for an individual participant. Flurpiridaz was administered on Study Day 1.
  Pharmacological stress agents were administered according to the respective Package Insert (as applicable) or American Society of Nuclear Cardiology or European Association of Cardiovascular Imaging standards corresponding to study site location.
- SPECT MPI: SPECT agents 99mTc-based myocardial tracers, example [99mTc]tetrofosmin or [99mTc]sestamibi were administered as per American Society of Nuclear Cardiology or European Association of Cardiovascular Imaging standards corresponding to study site location. For each participant, the same stress type (pharmacologic or exercise) was used for the SPECT and Flurpiridaz (18F) Injection PET MPI. Also, if pharmacological stress was used, the same agent and the same dose of pharmacological stress agent was used for both types of imaging for the same participant.
  Pharmacological stress agents were administered according to the respective Package Insert (as applicable) or American Society of Nuclear Cardiology or European Association of Cardiovascular Imaging standards corresponding to study site location.
Arm/Group | Flurpiridaz (18F) PET MPI | SPECT MPI
Number analyzed (Participants) | 578 | 578
percent
  Reader 1: Sensitivity: number analyzed (Participants) | 249 | 249
  Reader 1: Sensitivity | 77.1 [71.9 to 82.3] | 62.7 [56.6 to 68.7]
  Reader 1: Specificity: number analyzed (Participants) | 329 | 329
  Reader 1: Specificity | 65.7 [60.5 to 70.8] | 63.2 [58.0 to 68.4]
  Reader 2: Sensitivity: number analyzed (Participants) | 249 | 249
  Reader 2: Sensitivity | 73.5 [68.0 to 79.0] | 60.6 [54.6 to 66.7]
  Reader 2: Specificity: number analyzed (Participants) | 329 | 329
  Reader 2: Specificity | 69.6 [64.6 to 74.6] | 64.7 [59.6 to 69.9]
  Reader 3: Sensitivity: number analyzed (Participants) | 249 | 249
  Reader 3: Sensitivity | 88.8 [84.8 to 92.7] | 75.5 [70.2 to 80.8]
  Reader 3: Specificity: number analyzed (Participants) | 329 | 329
  Reader 3: Specificity | 52.6 [47.2 to 58.0] | 51.4 [46.0 to 56.8]
  Majority Rule: Sensitivity: number analyzed (Participants) | 249 | 249
  Majority Rule: Sensitivity | 80.3 [75.4 to 85.3] | 68.7 [62.9 to 74.4]
  Majority Rule: Specificity: number analyzed (Participants) | 329 | 329
  Majority Rule: Specificity | 63.8 [58.6 to 69.0] | 61.7 [56.4 to 67.0]
Statistical Analysis 1: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Reader 1: Sensitivity; Test type: Superiority — The test of sensitivity comparison between Flurpiridaz (18F) Injection PET MPI and SPECT MPI was performed with a 1-sided McNemar's test at a significance level of 0.025 using 1-sided McNemar's tests; p < 0.0001, McNemar; The hypothesis tests were 1-sided McNemar's tests with a significance level of 0.025 for sensitivity; Difference between PET MPI and SPECT MPI = 14.5, 95% CI 2-sided [6.5 to 22.4]
Statistical Analysis 2: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Reader 1: Specificity; Test type: Non-Inferiority — The test of specificity noninferiority between Flurpiridaz (18F) Injection PET MPI and SPECT MPI was performed with a paired test for noninferiority at a 1-sided significance level of 0.025 using Nam's RMLE method (margin=0.1); p = 0.0004, Nam's RMLE; Difference between PET MPI and SPECT MPI = 2.4, 95% CI 2-sided [-4.9 to 9.7]
Statistical Analysis 3: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Reader 2: Sensitivity; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0002, McNemar; Difference between PET MPI and SPECT MPI = 12.9, 95% CI 2-sided [4.7 to 21.0]
Statistical Analysis 4: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Reader 2: Specificity; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 2]; p < 0.0001, Nam's RMLE; Difference between PET MPI and SPECT MPI = 4.9, 95% CI 2-sided [-2.1 to 11.8]
Statistical Analysis 5: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Reader 3: Sensitivity; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, McNemar; Difference between PET MPI and SPECT MPI = 13.3, 95% CI 2-sided [6.6 to 19.9]
Statistical Analysis 6: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Reader 3: Specificity; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 2]; p = 0.0011, Nam's RMLE; Difference between PET MPI and SPECT MPI = 1.2, 95% CI 2-sided [-6.0 to 8.4]
Statistical Analysis 7: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Majority Rule: Sensitivity; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0003, McNemar; Difference between PET MPI and SPECT MPI = 11.6, 95% CI 2-sided [4.1 to 19.2]
Statistical Analysis 8: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Majority Rule: Specificity; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 2]; p = 0.0004, Nam's RMLE; Difference between PET MPI and SPECT MPI = 2.1, 95% CI 2-sided [-5.0 to 9.3]

3. Secondary Outcome: Sensitivity and Specificity of Flurpiridaz (18F) Injection PET MPI Compared SPECT MPI for Female Participants When the Diagnosis of CAD by ICA Was the Standard of Truth
Description: Sensitivity:TP/(TP+FN). TP:participants with abnormal PET MPI and disease positive by truth standard and FN:participants with normal PET MPI and disease positive by truth standard. Specificity:TN/(TN+ FP). TN:participants with normal PET MPI and disease negative by truth standard and FP:participants with abnormal PET MPI and disease negative by truth standard. Truth standard was presence of CAD as evidenced by presence of stenosis of >=50% in >=1 coronary artery or major branch of a coronary artery as determined by QCA analysis. Participants considered to have CAD if QCA revealed >=50% stenosis of >=1 major coronary artery or major branch. Sensitivity, specificity calculated for 3 readers and majority rule using each participant judgement (positive or negative) by at least 2 of 3 readers. Sensitivity, specificity of Flurpiridaz (18F) PET MPI compared to SPECT MPI with QCA as standard of truth at >=50% stenosis threshold for female participants was reported by reader and majority rule.
Time Frame: Up to 60 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Flurpiridaz (18F) PET MPI | SPECT MPI
Number analyzed (Participants) | 188 | 188
percent
  Reader 1: Sensitivity: number analyzed (Participants) | 41 | 41
  Reader 1: Sensitivity | 82.9 [71.4 to 94.4] | 58.5 [43.5 to 73.6]
  Reader 1: Specificity: number analyzed (Participants) | 147 | 147
  Reader 1: Specificity | 72.8 [65.6 to 80.0] | 63.3 [55.5 to 71.1]
  Reader 2: Sensitivity: number analyzed (Participants) | 41 | 41
  Reader 2: Sensitivity | 78.0 [65.4 to 90.7] | 56.1 [40.9 to 71.3]
  Reader 2: Specificity: number analyzed (Participants) | 147 | 147
  Reader 2: Specificity | 75.5 [68.6 to 82.5] | 68.7 [61.2 to 76.2]
  Reader 3: Sensitivity: number analyzed (Participants) | 41 | 41
  Reader 3: Sensitivity | 92.7 [84.7 to 100.0] | 75.6 [62.5 to 88.8]
  Reader 3: Specificity: number analyzed (Participants) | 147 | 147
  Reader 3: Specificity | 59.2 [51.2 to 67.1] | 58.5 [50.5 to 66.5]
  Majority Rule: Sensitivity: number analyzed (Participants) | 41 | 41
  Majority Rule: Sensitivity | 82.9 [71.4 to 94.4] | 65.9 [51.3 to 80.4]
  Majority Rule: Specificity: number analyzed (Participants) | 147 | 147
  Majority Rule: Specificity | 72.8 [65.6 to 80.0] | 66.0 [58.3 to 73.6]
Statistical Analysis 1: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Reader 1: Sensitivity; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0127, McNemar; Difference between PET MPI and SPECT MPI = 24.4, 95% CI 2-sided [5.4 to 43.4]
Statistical Analysis 2: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Reader 1: Specificity; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 2]; p = 0.0001, Nam's RMLE; Difference between PET MPI and SPECT MPI = 9.5, 95% CI 2-sided [-1.2 to 20.2]
Statistical Analysis 3: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Reader 2: Sensitivity; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0195, McNemar; Difference between PET MPI and SPECT MPI = 22.0, 95% CI 2-sided [2.2 to 41.7]
Statistical Analysis 4: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Reader 2: Specificity; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 2]; p = 0.0004, Nam's RMLE; Difference between PET MPI and SPECT MPI = 6.8, 95% CI 2-sided [-3.2 to 16.8]
Statistical Analysis 5: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Reader 3: Sensitivity; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0174, McNemar; Difference between PET MPI and SPECT MPI = 17.1, 95% CI 2-sided [1.7 to 32.4]
Statistical Analysis 6: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 2]; p = 0.0240, Nam's RMLE; Difference between PET MPI and SPECT MPI = 0.7, 95% CI 2-sided [-9.9 to 11.3]
Statistical Analysis 7: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Majority Rule: Sensitivity; Test type: Superiority; p = 0.0448, McNemar; Difference between PET MPI and SPECT MPI = 17.1, 95% CI 2-sided [-1.5 to 35.6]
Statistical Analysis 8: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Majority Rule: Specificity; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 2]; p = 0.0004, Nam's RMLE; Difference between PET MPI and SPECT MPI = 6.8, 95% CI 2-sided [-3.4 to 17.0]

4. Secondary Outcome: Sensitivity and Specificity of Flurpiridaz (18F) Injection PET MPI Compared SPECT MPI for Participants With Body-mass Index (BMI) >=30 Kilograms Per Square Meter (kg/m^2) When the Diagnosis of CAD by ICA Was the Standard of Truth
Description: Sensitivity:TP/(TP+FN). TP:participants with abnormal PET MPI and disease positive by truth standard and FN:participants with normal PET MPI and disease positive by truth standard. Specificity:TN/(TN+ FP). TN:participants with normal PET MPI and disease negative by truth standard and FP:participants with abnormal PET MPI and disease negative by truth standard. Truth standard was presence of CAD as evidenced by presence of stenosis of >=50% in >=1 coronary artery or major branch of coronary artery determined by QCA analysis. Participants considered to have CAD if QCA revealed >=50% stenosis of >=1 major coronary artery or major branch. Sensitivity, specificity calculated for 3 readers and majority rule using each participant judgement (positive or negative) by at least 2 of 3 readers. Sensitivity, specificity of Flurpiridaz (18F) PET MPI compared to SPECT MPI with QCA as standard of truth at >=50% stenosis threshold for participants(BMI>=30 kg/m^2) reported by reader and majority rule.
Time Frame: Up to 60 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Flurpiridaz (18F) PET MPI | SPECT MPI
Number analyzed (Participants) | 298 | 298
percent
  Reader 1: Sensitivity: number analyzed (Participants) | 117 | 117
  Reader 1: Sensitivity | 72.6 [64.6 to 80.7] | 60.7 [51.8 to 69.5]
  Reader 1: Specificity: number analyzed (Participants) | 181 | 181
  Reader 1: Specificity | 68.0 [61.2 to 74.8] | 61.3 [54.2 to 68.4]
  Reader 2: Sensitivity: number analyzed (Participants) | 117 | 117
  Reader 2: Sensitivity | 70.1 [61.8 to 78.4] | 63.2 [54.5 to 72.0]
  Reader 2: Specificity: number analyzed (Participants) | 181 | 181
  Reader 2: Specificity | 74.0 [67.6 to 80.4] | 62.4 [55.4 to 69.5]
  Reader 3: Sensitivity: number analyzed (Participants) | 117 | 117
  Reader 3: Sensitivity | 88.0 [82.2 to 93.9] | 74.4 [66.4 to 82.3]
  Reader 3: Specificity: number analyzed (Participants) | 181 | 181
  Reader 3: Specificity | 53.6 [46.3 to 60.9] | 50.8 [43.5 to 58.1]
  Majority Rule: Sensitivity: number analyzed (Participants) | 117 | 117
  Majority Rule: Sensitivity | 76.9 [69.3 to 84.6] | 69.2 [60.9 to 77.6]
  Majority Rule: Specificity: number analyzed (Participants) | 181 | 181
  Majority Rule: Specificity | 66.9 [60.0 to 73.7] | 61.9 [54.8 to 69.0]
Statistical Analysis 1: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Reader 1: Sensitivity; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0116, McNemar; Difference between PET MPI and SPECT MPI = 12.0, 95% CI 2-sided [0.0 to 23.9]
Statistical Analysis 2: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Reader 1: Specificity; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 2]; p = 0.0003, Nam's RMLE; Difference between PET MPI and SPECT MPI = 6.6, 95% CI 2-sided [-2.9 to 16.2]
Statistical Analysis 3: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Reader 2: Sensitivity; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.1085, McNemar; Difference between PET MPI and SPECT MPI = 6.8, 95% CI 2-sided [-5.2 to 18.9]
Statistical Analysis 4: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Reader 2: Specificity; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 2]; p < 0.0001, Nam's RMLE; Difference between PET MPI and SPECT MPI = 11.6, 95% CI 2-sided [2.1 to 21.1]
Statistical Analysis 5: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Reader 3: Sensitivity; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0017, McNemar; Difference between PET MPI and SPECT MPI = 13.7, 95% CI 2-sided [3.8 to 23.5]
Statistical Analysis 6: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Reader 3: Specificity; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 2]; p = 0.0034, Nam's RMLE; Difference between PET MPI and SPECT MPI = 2.8, 95% CI 2-sided [-6.6 to 12.1]
Statistical Analysis 7: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Majority Rule: Sensitivity; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0641, McNemar; Difference between PET MPI and SPECT MPI = 7.7, 95% CI 2-sided [-3.6 to 19.0]
Statistical Analysis 8: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Majority Rule: Specificity; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 2]; p = 0.0010, Nam's RMLE; Difference between PET MPI and SPECT MPI = 5.0, 95% CI 2-sided [-4.6 to 14.6]

5. Secondary Outcome: Sensitivity and Specificity of Flurpiridaz (18F) Injection PET MPI Compared SPECT MPI for Diabetic Participants When the Diagnosis of CAD by ICA Was the Standard of Truth
Description: Sensitivity:TP/(TP+FN). TP:participants with abnormal PET MPI and disease positive by truth standard and FN:participants with normal PET MPI and disease positive by truth standard. Specificity:TN/(TN+ FP). TN:participants with normal PET MPI and disease negative by truth standard and FP:participants with abnormal PET MPI and disease negative by truth standard. Truth standard was presence of CAD as evidenced by presence of stenosis of >=50% in >=1 coronary artery or major branch of coronary artery determined by QCA analysis. Participants considered to have CAD if QCA revealed >=50% stenosis of >=1 major coronary artery or major branch. Sensitivity and specificity calculated for 3 readers and majority rule using each participant judgement (positive or negative) by at least 2 of 3 readers. Sensitivity, specificity of Flurpiridaz (18F) PET MPI compared to SPECT MPI with QCA as standard of truth at >=50% stenosis threshold for diabetic participants was reported by reader and majority rule.
Time Frame: Up to 60 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Flurpiridaz (18F) PET MPI | SPECT MPI
Number analyzed (Participants) | 194 | 194
percent
  Reader 1: Sensitivity: number analyzed (Participants) | 91 | 91
  Reader 1: Sensitivity | 72.5 [63.4 to 81.7] | 61.5 [51.5 to 71.5]
  Reader 1: Specificity: number analyzed (Participants) | 103 | 103
  Reader 1: Specificity | 60.2 [50.7 to 69.6] | 56.3 [46.7 to 65.9]
  Reader 2: Sensitivity: number analyzed (Participants) | 91 | 91
  Reader 2: Sensitivity | 69.2 [59.7 to 78.7] | 62.6 [52.7 to 72.6]
  Reader 2: Specificity: number analyzed (Participants) | 103 | 103
  Reader 2: Specificity | 69.9 [61.0 to 78.8] | 58.3 [48.7 to 67.8]
  Reader 3: Sensitivity: number analyzed (Participants) | 91 | 91
  Reader 3: Sensitivity | 90.1 [84.0 to 96.2] | 81.3 [73.3 to 89.3]
  Reader 3: Specificity: number analyzed (Participants) | 103 | 103
  Reader 3: Specificity | 47.6 [37.9 to 57.2] | 39.8 [30.4 to 49.3]
  Majority Rule: Sensitivity: number analyzed (Participants) | 91 | 91
  Majority Rule: Sensitivity | 75.8 [67.0 to 84.6] | 71.4 [62.1 to 80.7]
  Majority Rule: Specificity: number analyzed (Participants) | 103 | 103
  Majority Rule: Specificity | 61.2 [51.8 to 70.6] | 51.5 [41.8 to 61.1]
Statistical Analysis 1: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Reader 1: Sensitivity; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0294, McNemar; Difference between PET MPI and SPECT MPI = 11.0, 95% CI 2-sided [-2.6 to 24.6]
Statistical Analysis 2: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Reader 1: Specificity; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 2]; p = 0.0117, Nam's RMLE; Difference between PET MPI and SPECT MPI = 3.9, 95% CI 2-sided [-8.3 to 16.1]
Statistical Analysis 3: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Reader 2: Sensitivity; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.1444, McNemar; Difference between PET MPI and SPECT MPI = 6.6, 95% CI 2-sided [-7.1 to 20.3]
Statistical Analysis 4: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Reader 2: Specificity; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 2]; p = 0.0001, Nam's RMLE; Difference between PET MPI and SPECT MPI = 11.7, 95% CI 2-sided [-0.4 to 23.7]
Statistical Analysis 5: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Reader 3: Sensitivity; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0440, McNemar; Difference between PET MPI and SPECT MPI = 8.8, 95% CI 2-sided [-1.3 to 18.9]
Statistical Analysis 6: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Reader 3: Specificity; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 2]; p = 0.0022, Nam's RMLE; Difference between PET MPI and SPECT MPI = 7.8, 95% CI 2-sided [-4.8 to 20.3]
Statistical Analysis 7: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Majority Rule: Sensitivity; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.2164, McNemar; Difference between PET MPI and SPECT MPI = 4.4, 95% CI 2-sided [-8.4 to 17.2]
Statistical Analysis 8: Comparison: Flurpiridaz (18F) PET MPI vs SPECT MPI; Majority Rule: Specificity; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 2]; p = 0.0006, Nam's RMLE; Difference between PET MPI and SPECT MPI = 9.7, 95% CI 2-sided [-2.6 to 22.0]

ADVERSE EVENTS:
Time Frame: From the time of informed consent to end of follow up (up to 77 days)
Description: The Safety population consisted of all enrolled participants who received >=1 dose of Flurpiridaz (18F) Injection in the study.
Groups:
- Flurpiridaz (18F): Safety Population: Participants received 2 IV boluses of Flurpiridaz (18F) Injection in a large peripheral vein: 1 at rest then 1 during stress on the same day within 60 days prior to the ICA. Flurpiridaz (18F) Injection administered at rest and during stress conditions were not to exceed a total of 14 mCi (520 MBq) for an individual participant. Flurpiridaz was administered on Study Day 1.
  SPECT agents 99mTc-based myocardial tracers, example [99mTc]tetrofosmin or [99mTc]sestamibi were administered as per American Society of Nuclear Cardiology or European Association of Cardiovascular Imaging standards corresponding to study site location. For each participant, the same stress type (pharmacologic or exercise) was used for the SPECT and Flurpiridaz (18F) Injection PET MPI. Also, if pharmacological stress was used, the same agent and the same dose of pharmacological stress agent was used for both types of imaging for the same participant.
  Pharmacological stress agents were administered according to the respective Package Insert (as applicable) or American Society of Nuclear Cardiology or European Association of Cardiovascular Imaging standards corresponding to study site location.
Arm/Group | Flurpiridaz (18F): Safety Population
All-Cause Mortality (participants affected / at risk) | 1/604
Serious Adverse Events (participants affected / at risk) | 20/604
Other Adverse Events (participants affected / at risk) | 145/604
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Flurpiridaz (18F): Safety Population (N=604)
Acute myocardial infarction (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 2
Angina unstable (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Coronary artery perforation (Cardiac disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Chest pain (General disorders) | 1
Vascular stent thrombosis (General disorders) | 1
Anaphylactic shock (Immune system disorders) | 1
Post procedural fever (Injury, poisoning and procedural complications) | 1
Electrocardiogram abnormal (Investigations) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Urticaria chronic (Skin and subcutaneous tissue disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Flurpiridaz (18F): Safety Population (N=604)
Angina pectoris (Cardiac disorders) | 32
Headache (Nervous system disorders) | 80
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI and/or institution is that the Sponsor can review results communications prior to public release and can restrict communications regarding trial results for a period that is more than 30 days (publications/abstracts) but not to exceed 90 days (patent related issues) from the time submitted to the Sponsor to review. The PI may be asked to remove any Sponsor confidential information and/or delay publication to protect any proprietary information.

DOCUMENTS (2):
  • Study Protocol (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT03354273/Prot_002.pdf
  • Statistical Analysis Plan (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT03354273/SAP_003.pdf